CLINICAL TRIAL: NCT01486186
Title: Detection and Intervention on Mild/Moderate Chronic Obstructive Pulmonary Disease by Traditional Chinese Medicine Treatment and Application
Brief Title: Effect of Traditional Chinese Medicine on Outcomes in Patients With Mild/Moderate Chronic Obstructive Pulmonary Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Henan University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TCM for COPD
Record Dates: First submitted 2011-11-15; First posted 2011-12-06 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2011-12

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Pulmonary Disease, Chronic Obstructive; Double-Blind Method; Medicine, Chinese Traditional; Humans; Treatment Outcome
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Medicine, Chinese Traditional

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- traditional chinese medicine (Experimental): The experimental group will receive three type of TCM, they are Baofei granule, Bufeijianpi granule and Bufeiyishen granule.
  Interventions: Drug: Traditional Chinese Medicine
- placebo (Placebo Comparator): placebo chinese medicine in addition to best care according to clinical guidelines for COPD patients
  Interventions: Drug: placebo chinese medicine

INTERVENTIONS:
Drug: Traditional Chinese Medicine — A herbal extract twice daily for 52 weeks for lower dosage, There are 3 Recipe for the 3 traditional Chinese syndrome, they are syndrome of lung-qi deficiency, syndrome of deficiency of pulmonosplenic qi, syndrome of insufficiency of QI of the lung and kidney.
  Other Names: Baofei granule; Bufeijianpi granule; Bufeiyishen granule
  Arms: traditional chinese medicine
Drug: placebo chinese medicine — There are 3 placebo Recipe for the 3 traditional Chinese syndrome.
  Other Names: placebo Baofei granule; placebo Bufeijianpi granule; placebo Bufeiyishen granule
  Arms: placebo

SUMMARY:
The purpose of this study is evaluate the effects and safety of Traditional Chinese medicine for prevention and management of mild/moderate chronic obstructive pulmonary disease (COPD).

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo controlled study to evaluate the effect of Traditional Chinese medicine (TCM) in COPD subjects. Following a 14 day run-in period, approximately 504 subjects will be randomly assigned to double-blind treatment for 52 weeks. After the 52 weeks treatment period, subjects in both treatment arms will follow-up 52 weeks. The primary measure of efficacy is the frequency of exacerbations and spirometric values (e.g. FEV1). Secondary efficacy measures include Dyspnea (MMRC), Quality of life ( CAT,SF-36), Exercise Capacity( 6MWD). Safety will be assessed through the collection of adverse events. There will be a total of 5 study visits ( randomization, and after 13, 26, 39 and 52 weeks of treatment). A follow-up contact for collection of effect and adverse event will be conducted approximately 52 weeks following the last study visit.

ELIGIBILITY:
Inclusion Criteria:

* A confirmed diagnosis of mild/moderate COPD.
* Age between 40 and 80 years.
* Syndrome differentiation belongs to Syndrome of lung-qi deficiency, Syndrome of deficiency of pulmonosplenic qi, Syndrome of insufficiency of QI of the lung and kidney.
* Without participation in other interventional trials in the previous one month.
* With the informed consent signed.

Exclusion Criteria:

* Pregnant or breast-feeding women.
* Any psychiatric condition rendering the patient unable to understand the nature, scope and possible consequences of the study .
* Complicated with severe heart failure (class Ⅳ NYHA heart function) or unstable hemodynamics.
* Complicated with bronchial asthma, bronchiectasis or active tuberculosis；
* Complicated with obliterative bronchiolitis or diffuse pantothenic bronchiolitis，
* Complicated with pneumothorax, pleural effusion or pulmonary embolism.
* Complicated with neuromuscular disorder which affects the respiration.
* Complicated with tumors.
* Complicated with serious hepatic and renal diseases.
* Long periods of bed rest.
* Use of oral or parenteral corticosteroids before 1 months of Visit 1 .
* With immunodeficiency.
* Participating in other trials or allergic to the used medicine.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 504 (Estimated)
Dates: Start 2011-12; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
pulmonary function（FEV1） | Change from Baseline in FEV1 at Week 26 and 52 of the treatment phase, Week 26 and 52 of the followup phase
the frequency of exacerbation | Change from Baseline in the frequency of exacerbation at Week 26 and 52 of the treatment phase, Week 26 and 52 of the followup phase

SECONDARY OUTCOMES:
Dyspnea | Change from Baseline in MMRC at Week 13, 26, 39 and 52 of the treatment phase, Week 26 and 52 of the followup phase
Quality of life | Change from Baseline in CAT and SF-36 at Week 13, 26, 39 and 52 of the treatment phase, Week 26 and 52 of the followup phase
  using COPD Assessment Test ( CAT) and short-form 36-item questionnaire (SF-36)
6 Minutes Walking Distance Test ( 6MWD) | Change from Baseline in 6MWD at Week 13, 26, 39 and 52 of the treatment phase, Week 26 and 52 of the followup phase

CONTACTS AND LOCATIONS:
Overall Officials: Li jiansheng, doctor, Study Chair — The First Affiliated Hospital of Henan University of Traditional Chinese Medicine

REFERENCES:
- [Derived] Wang M, Li J, Li S, Wang H, Yu X, Zhang H. Effect of traditional Chinese medicine on outcomes in patients with mild/moderate chronic obstructive pulmonary disease: study protocol for a randomized placebo-controlled trial. Trials. 2012 Jul 16;13:109. doi: 10.1186/1745-6215-13-109. PMID 22799753